CLINICAL TRIAL: NCT04437420
Title: Preclinical Project on the Traitment of Acute Lymphoblastique Leukemia With NVP-BEP800, an Inhibitor of the Heat Shock Protein HSP90
Acronym: HSP-HEMATO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: GIRODON Collection 2020
Record Dates: First submitted 2020-06-16; First posted 2020-06-18 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Acute T Lymphoblastic Leukemia (T-ALL); Acute B Lymphoblastic Leukemia (B-ALL)
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- T-ALL
  Interventions: Drug: injection of BEP 800; Other: Control
- B-ALL
  Interventions: Drug: injection of BEP 800; Other: Control

INTERVENTIONS:
Drug: injection of BEP 800 — injection of BEP 800
Other: Control — no injection of BEP 800

SUMMARY:
NVP-BEP800, a new HSP90 inhibitor, has particularly interesting therapeutic potential and represents hope in cancer pathologies. While it is currently being tested for solid cancers, no preclinical study has yet demonstrated its effectiveness in acute lymphoblastique leukemia (ALL). The investigators wish to study the effects of NVP-BEP800 on two different types of ALL (T and B-ALL).

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering from acute lymphoblastic leukaemia whose biological samples are kept at the Biology Technical Platform.

Exclusion Criteria:

* Patient over 80 years of age

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with acute lymphoblastic leukemia with biological samples stored at the Biology Technical Platform.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Viability on primary ALL samples | 2 years
  The effect of BEP-800 after 48 hours of treatment on T-ALL and B-ALL will be evaluated by counting viable cells by flow cytometry with a viability marker and specific antibodies to detect leukemia cells.

SECONDARY OUTCOMES:
Effect on SRC phosphorylation | 2 years
  The effect of BEP-800 on T-ALL and B-ALL will be evaluated by flow cytometry by measuring HSP90 and SRC (phosphorylated), by intracellular labeling after permeabilization of the cells, 18 hours after treatment with BEP-800.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France